CLINICAL TRIAL: NCT04399330
Title: Hypermobility and Obstructions in the Craniocervical Region Among Patients With Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
Brief Title: ME/CFS, Hypermobility and Craniocervical Obstructions
Status: Completed | Type: Observational
Sponsor: Bragee Clinics (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: Meret2019
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective study on clinical and radiological findings in ME/CFS

ELIGIBILITY:
Inclusion Criteria:

Patients at a multidisciplinary specialist clinic accepting to participate

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 190 women 39 men Mean duration 9 years
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of cervical obstruction and other MRI findings | 1990-2020
  Findings as disc bulging, disc hernias, chiari malformations
Prevalence of hypermobility | 1990-2020
  Measured as Beighton score and other signs of Ehlers Danlos syndrome (EDS) variations

CONTACTS AND LOCATIONS:
Overall Officials: Björn Bragée, MD, Study Director — Bragee Clinics
Locations (1):
- Bragee Clinics, Stockholm, Sweden